CLINICAL TRIAL: NCT04470479
Title: Oral Pilocarpine in the Treatment of the Dry Eye of Patients With Sjogrens Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Sergio Felberg, Posgraduate Medical Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0910/03
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye
Keywords: dry eye; Sjogren; pilocarpine hydrochloride
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Pilocarpine

STUDY DESIGN:
Intervention Model Description: This was a placebo-controlled, crossover study that involved patients with Sjögren's syndrome to use 20mg/day of oral pilocarpine or placebo for ten weeks and after two weeks of medication withdrawal, to invert the treatment for the same period of time. The assessments applied were the Ocular Surface Disease Index, NEI-VFQ-25 questionnaire, non-invasive break-up time, traditional break-up time, evaluation of the cornea and ocular surface with fluorescein and rose bengal dyes, Schirmer test, tear ferning test, osmolarity and the activity of lysozyme. R
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pilocarpine Hydrochloride (Experimental): Patients with Sjögren's syndrome were allocated to receive oral pilocarpine 20mg per day, (5mg every 6 hours, for ten weeks.
  Interventions: Drug: Pilocarpine Hydrochloride
- placebo (Placebo Comparator): Patients with Sjögren's syndrome were allocated to receive placebo administered in the same way (1 tablet every 6 hours), for ten weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pilocarpine Hydrochloride — Oral pilocarpine hydrochloride 5mg tablets were administered four times a day for 10 weeks to half the group of selected patients. The other half ingested placebo in the same way. At the end of this period and after two weeks of washing out the medications, the patients had to invert the treatments.
  Other Names: Salagen
  Arms: Pilocarpine Hydrochloride
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
The purpose of this study was to access the possible beneficial effects of oral use of pilocarpine in relieving signs and symptoms of patients with Sjogren's syndrome

DETAILED DESCRIPTION:
After being informed about the study, its potential risks and having signed the informed consent form, this placebo-controlled, crossover study involved patients with Sjögren's syndrome to use oral pilocarpine or placebo for ten weeks and after two weeks of medication withdrawal, to invert the treatment for the same period of time. The assessments applied were the Ocular Surface Disease Index, NEI-VFQ-25 questionnaire, non-invasive break-up time, traditional break-up time, evaluation of the cornea and ocular surface with fluorescein and rose bengal dyes, Schirmer test, and tear ferning test. Side effects observed during the treatment period were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sjögren's syndrome, both in primary and secondary forms, whose diagnoses were established according to the criteria defined by the - American-European Consensus for the diagnosis of Sjögren's syndrome.
* Patients with the secondary form of the syndrome, collagen disease considered controlled by a rheumatologist, before the start of the trial and stable until the end of the study.
* Systemic therapy instituted up to two months before the beginning of the protocol.
* Literate patients.
* Signature of the informed consent form

Exclusion Criteria:

* Eye or eyelid surface disease not attributed to Sjogren's syndrome.
* Temporary or permanent occlusion of tear points.
* Use of contact lenses.
* Use of systemic medication that is known to influence tear flow.
* Need to modify the systemic treatment of the underlying disease during the trial.
* Pregnancy or breastfeeding.
* Known hypersensitivity reaction to pilocarpine hydrochloride.
* Severe cardio-pulmonary disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2006-04-01 (Actual); Study Completion 2006-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Ocular Surface Disease Index questionnaire at week 10 | Baseline and week 10
  The Ocular Surface Disease Index is a valid and reliable instrument for measuring the severity of dry eye disease, and it possesses the necessary psychometric properties to be used as an end point in clinical trials. The answers to the questions generate an index ranging from 0 to 100, where 0 means no complaints related to dry eye and 100 indicates complaints with maximum intensity. (Change = week 10 score - baseline score)
Change from baseline Ocular Surface Disease Index questionnaire at week 22 | Baseline and week 22
  The Ocular Surface Disease is a valid and reliable instrument for measuring the severity of dry eye disease, and it possesses the necessary psychometric properties to be used as an end point in clinical trials. The answers to the questions generate an index ranging from 0 to 100, where 0 means no complaints related to dry eye and 100 indicates complaints with maximum intensity. (Change = week 22 score - baseline score)
Change from baseline in the NEI-VFQ-25 questionnaire at week 10 | Baseline and week 10
  The VFQ-25 is a reliable and validated 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration. The set of responses provided scores between 0 and 100, where 0 means the maximum negative impact of the disease on the quality of life of patients and 100 means no negative impact of the disease on quality of life. (Change = week 10 score - baseline score)
Change from baseline in the NEI-VFQ-25 questionnaire at week 22 | Baseline and week 22
  The VFQ-25 is a reliable and validated 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration. The set of responses provided scores between 0 and 100, where 0 means the maximum negative impact of the disease on the quality of life of patients and 100 means no negative impact of the disease on quality of life. (Change = week 22 score - baseline score)
Change from baseline in tear breakup time test at week 10 | Baseline and week 10
  Tear breakup time is a clinical test used to assess evaporative disease of dry eye. To measure tear breakup time, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is viewed under a cobalt blue lighting. The time of appearance of the first tear film break point, recorded in seconds, indicates the tear film breakup time. Times greater than 10 seconds are considered normal. (Change = week 10 measure - baseline measure)
Change from baseline in tear breakup time test at week 22 | Baseline and week 22
  Tear breakup time is a clinical test used to assess evaporative disease of dry eye. To measure tear breakup time, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is viewed under a cobalt blue lighting. The time of appearance of the first tear film break point, recorded in seconds, indicates the tear film breakup time. Times greater than 10 seconds are considered normal. (Change = week 22 measure - baseline measure)
Change from baseline in score with rose bengal staining at week 10 | Baseline and week 10
  When instilled in the ocular surface, the rose bengal dye will stain dead cells and spaces not covered by the tear film, being a method used to evaluate the damage to the ocular surface caused by the dry eye. For quantification, the van bijesterveld scale was used, which gives a score from 0 to 9 points according to the intensity of the color distributed onto the ocular surface. The van bijesterveld scale is described as follows:
  The surface of the eye should be separated into three regions: the nasal bulbar conjunctiva, the cornea and the medial bulbar conjunctiva. Each of these regions may receive a score ranging from 0 to 3 points (0 = not colored, 1 = colored with distant points, 2 = colored with close points and 3 = colored with confluent points). The scores are then added up, generating a global score ranging from 0 to 9 points. Score 0 means no impairment of the ocular surface and score 9 means maximum impairment of the ocular surface).
  (Change = week 10 - baseline measure)
Change from baseline in score with rose bengal staining at week 22 | Baseline and week 22
  When instilled in the ocular surface, the rose bengal dye will stain dead cells and spaces not covered by the tear film, being a method used to evaluate the damage to the ocular surface caused by the dry eye. For quantification, the van bijesterveld scale was used, which gives a score from 0 to 9 points according to the intensity of the color distributed onto the ocular surface. The van bijesterveld scale is described as follows:
  The surface of the eye should be separated into three regions: the nasal bulbar conjunctiva, the cornea and the medial bulbar conjunctiva. Each of these regions may receive a score ranging from 0 to 3 points (0 = not colored, 1 = colored with distant points, 2 = colored with close points and 3 = colored with confluent points). The scores are then added up, generating a global score ranging from 0 to 9 points. Score 0 means no impairment of the ocular surface and score 9 means maximum impairment of the ocular surface).
  (Change = week 22 - baseline measure)
Change from baseline in corneal keratitis score with fluorescein dye at week 10 | Baseline and week 10
  After dripping fluorescein dye on the ocular surface, the cornea of the patients was analyzed with the patient accommodated in the slit lamp and under cobalt blue light. Fluorescein will stain spaces without cells, which represents spaces in distress caused by dry eyes. The score used ranges from 0 to 3 points (0 = not colored, 1 = blush with distant points, 2 = blush with close points and 3 = blush with confluent points). Score 0 means no corneal involvement (absence of keratitis) and score 3 means maximum involvement of the ocular surface) (Change = week 10 - baseline score)
Change from baseline in corneal keratitis score with fluorescein dye at week 22 | Baseline and week 22
  After dripping fluorescein dye on the ocular surface, the cornea of the patients was analyzed with the patient accommodated in the slit lamp and under cobalt blue light. Fluorescein will stain spaces without cells, which represents spaces in distress caused by dry eyes. The score used ranges from 0 to 3 points (0 = not colored, 1 = blush with distant points, 2 = blush with close points and 3 = blush with confluent points). Score 0 means no corneal involvement (absence of keratitis) and score 3 means maximum involvement of the ocular surface) (Change = week 22 - baseline score)
Change from baseline in The Schirmer test at week 10 | Baseline and week 10
  The Schirmer test measures, in millimeters, the production of the tear film for five minutes. A strip of standardized paper is placed on the lateral third of the lower eyelid of both eyes and after 5 minutes. The tear moistens the paper and the reading of the moistening is done. The test can vary from 0 to 35 millimeters, being considered normal (normal tear flow) values greater than 10 millimeters. Values below 10 millimeters indicate dry eye and the lower the value, the more dry the eye.
  (Change = week 10 - baseline measure)
Change from baseline in The Schirmer test at week 22 | Baseline and week 22
  The Schirmer test measures, in millimeters, the production of the tear film for five minutes. A strip of standardized paper is placed on the lateral third of the lower eyelid of both eyes and after 5 minutes. The tear moistens the paper and the reading of the moistening is done. The test can vary from 0 to 35 millimeters, being considered normal (normal tear flow) values greater than 10 millimeters. Values below 10 millimeters indicate dry eye and the lower the value, the more dry the eye.
  (Change = week 22 - baseline measure)
Change from baseline in Tear ferning test (Rolando'score) at week 10 | Baseline and week 10
  The tear ferning test is a laboratory test but it has the potential to be applied in the clinic setting to investigate the tear film in a simple way. Drying a small sample of tear fluid onto a clean, glass microscope slide produces a characteristic crystallisation pattern, described as a 'tear ferning". The scale proposed by Rolando was used, which classifies the findings into 4 types (type 1, 2, 3 and 4), according to the teardrop crystallization pattern. Patterns 1 and 2 are considered normal and patterns 3 and 4 are considered abnormal and indicate that the tear has an inadequate composition and quality (Change = week 10 - baseline score)
Change from baseline in Tear ferning test (Rolando'score) at week 22 | Baseline and week 22
  The tear ferning test is a laboratory test but it has the potential to be applied in the clinic setting to investigate the tear film in a simple way. Drying a small sample of tear fluid onto a clean, glass microscope slide produces a characteristic crystallisation pattern, described as a 'tear ferning". The scale proposed by Rolando was used, which classifies the findings into 4 types (type 1, 2, 3 and 4), according to the teardrop crystallization pattern. Patterns 1 and 2 are considered normal and patterns 3 and 4 are considered abnormal and indicate that the tear has an inadequate composition and quality (Change = week 22 - baseline score)

SECONDARY OUTCOMES:
The frequency of systemic side effects most frequently reported by patients at week 10 | week 10
  A list of the systemic side effects most frequently described with the oral use of pilocarpine was presented to patients, where they could indicate the presence or absence of this effect: the side effects on the list are: sweating, chills, nausea, salivation, abdominal pain, dizziness, facial flushing, rhinitis, weakness, visual blurring, tremor, tachycardia, headache and diarrhea.
The frequency of systemic side effects most frequently reported by patients at week 22 | week 22
  A list of the systemic side effects most frequently described with the oral use of pilocarpine was presented to patients, where they could indicate the presence or absence of this effect: the side effects on the list are: sweating, chills, nausea, salivation, abdominal pain, dizziness, facial flushing, rhinitis, weakness, visual blurring, tremor, tachycardia, headache and diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Felberg, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Irmandade Santa casa de Misericórdia de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Detailed description of the methods may be made available after publication
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication, for 3 months
Access Criteria: IPD may be requested from the principal investigator upon request by email or letter addressed to registered contacts

REFERENCES:
- [Result] Kawakita T, Shimmura S, Tsubota K. Effect of Oral Pilocarpine in Treating Severe Dry Eye in Patients With Sjogren Syndrome. Asia Pac J Ophthalmol (Phila). 2015 Mar-Apr;4(2):101-5. doi: 10.1097/APO.0000000000000040. PMID 26065354
- [Result] Cifuentes M, Del Barrio-Diaz P, Vera-Kellet C. Pilocarpine and artificial saliva for the treatment of xerostomia and xerophthalmia in Sjogren syndrome: a double-blind randomized controlled trial. Br J Dermatol. 2018 Nov;179(5):1056-1061. doi: 10.1111/bjd.16442. Epub 2018 May 29. PMID 29432648
- [Result] Papas AS, Sherrer YS, Charney M, Golden HE, Medsger TA Jr, Walsh BT, Trivedi M, Goldlust B, Gallagher SC. Successful Treatment of Dry Mouth and Dry Eye Symptoms in Sjogren's Syndrome Patients With Oral Pilocarpine: A Randomized, Placebo-Controlled, Dose-Adjustment Study. J Clin Rheumatol. 2004 Aug;10(4):169-77. doi: 10.1097/01.rhu.0000135553.08057.21. PMID 17043506